CLINICAL TRIAL: NCT05426733
Title: An Open-label Extension Study to Evaluate Long-term Efficacy and Safety of Odevixibat (A4250) in Children With Biliary Atresia (BOLD-EXT)
Brief Title: An Open-label Extension Study to Evaluate Long-term Efficacy and Safety of Odevixibat in Children With Biliary Atresia
Acronym: BOLD-EXT
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Albireo, an Ipsen Company (Industry)
Responsible Party: Sponsor
Organization: Ipsen (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A4250-016; 2022-501090-39-00 (EU CTIS Number)
Record Dates: First submitted 2022-06-13; First posted 2022-06-22 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Biliary Atresia
MeSH Terms: conditions — Biliary Atresia | interventions — odevixibat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Odevixibat (A4250) (Experimental): Capsules for oral administration once daily for 104 weeks.
  Interventions: Drug: Odevixibat

INTERVENTIONS:
Drug: Odevixibat — Odevixibat is a small molecule inhibitor of the ileal bile acid transporter (IBAT).
  Other Names: A4250

SUMMARY:
An Open-label Extension Study to Evaluate Long-term Efficacy and Safety of Odevixibat (A4250) in Children with Biliary Atresia

DETAILED DESCRIPTION:
This is a Phase 3, multi-center, open-label extension study to evaluate the long-term efficacy and safety of odevixibat in patients with Biliary Atresia (BA). Patients who completed treatment in the A4250-011 BOLD study and meet eligibility criteria for Study A4250-016 (BOLD-EXT) can participate. The duration of the treatment period is 104 weeks, followed by a 4-week Safety Follow-up Period. Patients who wish to continue receiving odevixibat after 104 weeks can remain on treatment in the optional extension period (OEP).

Up to 180 patients will be enrolled at approximately 70 sites in the North America, Europe, the Middle East and Asia-Pacific.

ELIGIBILITY:
Inclusion Criteria:

* Completion of the 104-week Treatment Period of Study A4250-011
* Signed informed consent by caregiver

Exclusion Criteria:

* Patients who were not compliant with study drug treatment or procedures in Study A4250-011 as per the investigator's discretion
* Any conditions or abnormalities which, in the opinion of the investigator, may compromise the safety of the patient, or interfere with the patient participating in or completing the study
* Known hypersensitivity to any components of odevixibat
* Patients who are scheduled for a liver transplant or are likely to require a liver transplant in the immediate future based on the investigator's judgment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-07-05 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who are alive and have not undergone liver transplant | From baseline to Week 104

SECONDARY OUTCOMES:
Change in aspartate aminotransferase (AST) to platelet ratio index (APRI) score | From baseline to Week 104
  The APRI (aspartate aminotransferase to platelet ratio index) score estimates the severity of liver fibrosis. A higher score indicates a greater amount of scarring (fibrosis) in the liver.
  * A score ≤ 0.5 indicates a low likelihood of fibrosis
  * A score ≥ 1.5 indicates a higher probability of fibrosis
Change in Fibrosis-4 (Fib-4) score | From baseline to Week 104
  The Fib-4 score provides an estimate of the amount of scarring (fibrosis) in the liver. A higher score indicates a greater amount of scarring in the liver.
  * A score < 1.45 indicates a low likelihood of fibrosis
  * A score > 3.25 indicates a higher probability of fibrosis
Change in serum bile acids | From Baseline to Weeks 26, 52, 78, and 104
Change in height | From Baseline to Weeks 26, 52, 78 and 104
Change in weight | From Baseline to Weeks 26, 52, 78 and 104
Change in mid-arm circumference | From Baseline to Weeks 26, 52, 78 and 104
  Measure of growth
Time to onset of any sentinel events | From Baseline to Week 104
Change in pediatric end-stage liver disease (PELD) score | From Baseline to Weeks 26, 52, 78 and 104
  The PELD (pediatric end-stage liver disease) score is a measure of disease severity. PELD scores can range from a negative value (such as -10) to high numbers (such as 45). A higher score indicates more severe disease.

CONTACTS AND LOCATIONS:
Locations (30):
- United States (10):
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's Healhcare of Atlanta- Emory University school of medicine, Atlanta, Georgia
  - Indiana University school of Medicine, Indianapolis, Indiana
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Mercy Hospital and Clinics, Kansas City, Missouri
  - Hassenfeld Children's Hospital at NYU Langone, New York, New York
  - Columbia University Medical Center New York Presbyterian Morgan Stanley-Komansky Childrens Hospital, New York, New York
  - The Childrens Hospital at Montefiore Albert Einstein School of Medicine, The Bronx, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Seattle Children's Hospital, Seattle, Washington
- Royal Children's Hospital, Parkville, Australia
- Canada (2):
  - CHU Sainte-Justine, Montreal
  - The Hospital for Sick Children, Toronto
- China (2):
  - Guangzhou Women And Childrens Medical Center, Guangdong
  - Children's Hospital of Fudan University, Shanghai
- Bicêtre Hospital, Le Kremlin-Bicêtre, France
- Germany (2):
  - Charité - Universitätsmedizin Berlin, Berlin
  - University Children´s Hospital Tuebingen, Tübingen
- Italy (2):
  - ASST Papa Giovanni XXIII, Bergamo
  - Azienda Ospedaliera di Padova, Padua
- Malaysia (2):
  - Hospital Raja Perempuan Zainab II, Kota Bharu
  - University Malaya Medical Centre, Kuala Lumpur
- University Medical Center Groningen, Groningen, Netherlands
- Starship Child Health, Te Whatu Ora - Health New Zealand, Auckland, New Zealand
- Instytut Pomnik-Centrum Zdrowia Dziecka, Warsaw, Poland
- Seoul National University Childrens Hospital, Seoul, South Korea
- Hospital Universitari Vall d'Hebron, Barcelona, Spain
- Turkey (Türkiye) (3):
  - Hacettepe İhsan Doğramacı Children's Hospital, Ankara
  - Akdeniz University Medical Faculty, Antalya
  - Istanbul University Istanbul Medical Faculty Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications.
  Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and/or EU.
Access Criteria: Further details on Ipsen's sharing criteria and process for sharing are available here (https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/).
URL: https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/